CLINICAL TRIAL: NCT02001506
Title: A Randomized Phase III Trial of Neoadjuvant Chemotherapy With 3 Cycles of FEC Followed by 3 Cycles of Docetaxel Versus 4 Cycles of Adriamycin Plus Cyclophosphamide Followed by 4 Cycles of Docetaxel in Node-positive Breast Cancer
Brief Title: Neoadjuvant Chemotherapy of 6 Cycles vs 8 Cycles in Node Positve Breast Cancer
Acronym: Neo-shorter
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Bae Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0116
Record Dates: First submitted 2013-11-19; First posted 2013-12-05 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; neoadjuvant; different number of chemotherapy cycles
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorouracil; Epirubicin; Cyclophosphamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FEC3-D3 (Active Comparator): 3 cycles of FEC followed by 3 cycles of Docetaxel
  Fluorouracil 500 mg/m2, every 3 weeks Epirubicin 100 mg/m2, every 3 weeks Cyclophosphamide 500, every 3 weeks
  Docetaxel 75 mg/m2, every 3 weeks
  Interventions: Drug: FEC3-D3
- AC4-D4 (No Intervention): 4 cycles of Adriamycin plus Cyclophosphamide (AC) followed by 4 cycles of Docetaxel
  Adriamycin 60 mg/m2, every 3 weeks Cyclophosphamide 600 mg/m2, every 3 weeks
  Docetaxel 75 mg/m2, every 3 weeks

INTERVENTIONS:
Drug: FEC3-D3 — Fluorouracil 500 mg/m2, every 3 weeks Epirubicin 100 mg/m2, every 3 weeks Cyclophosphamide 500, every 3 weeks
  Docetaxel 75 mg/m2, every 3 weeks
  Other Names: 5-FU; Pharmorubicin; Cytoxan; Docetaxel
  Arms: FEC3-D3

SUMMARY:
Various regimens and schedule as neoadjuvant chemotherapy regimens were investigated and sequential treatment of anthracyclines followed by taxanes, which has shown superior pathologic complete respone (pCR) rate (NSABP-B27 study) is widely used until now. Considering the proven efficacy and tolerable toxicity of 3 cycles of FEC followed by 3 cycles of Docetaxel (FEC3-D3) compared to FEC 6 cycles in adjuvant chemotherapy (PACS 01 trial), use of FEC3-D3 regimen in neoadjuvant setting will be feasible with acceptable efficacy and further reduce the duration of neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
To investigate feasibility of FEC3-D3 regimen in neoadjuvant setting in terms of comparable efficacy and shorter duration across all subtypes.

ELIGIBILITY:
Inclusion Criteria:

* Performance status 0 or 1
* Clinically stage 2 or 3 with histologically proven lymph node involvement
* Tumor or lymph node greater than 1.5 cm

Exclusion Criteria:

* Pregnancy or lactation
* Prior chemotherapy or radiotherapy for any malignancy
* Documented history of cardiac disease contraindicating anthracyclines
* Currently active infection

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2012-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
pathologic complete response (pCR) between two arms | within the first 30 days (plus or minus 3 days) after surgery

SECONDARY OUTCOMES:
3 year-disease free survival between two arms | 3 year after surgery
  1. Correlation of pCR and Ki-67 expression at baseline and D14 tumor specimen
  2. 3 year-disease free survival
  3. Correlation of pCR and biomarkers such as Ki-67 expression

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Bae Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Hwang I, Kim JE, Jeong JH, Ahn JH, Jung KH, Son BH, Kim HH, Shin J, Lee HJ, Gong G, Kim SB. Randomized phase III trial of a neoadjuvant regimen of four cycles of adriamycin plus cyclophosphamide followed by four cycles of docetaxel (AC4-D4) versus a shorter treatment of three cycles of FEC followed by three cycles of docetaxel (FEC3-D3) in node-positive breast cancer (Neo-shorter; NCT02001506). Breast Cancer Res Treat. 2023 Sep;201(2):193-204. doi: 10.1007/s10549-023-06971-7. Epub 2023 Jun 26. PMID 37365483